CLINICAL TRIAL: NCT04929613
Title: Intensive Mindfulness-based Resilience Training in First Responders: A Pilot Study
Brief Title: Resilience Training for First Responders in the Opioid Epidemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1704554931
Record Dates: First submitted 2021-06-02; First posted 2021-06-18 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Compassion Fatigue; Burnout; Stress; Mindfulness
Keywords: First Responders
MeSH Terms: conditions — Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Resilience Training (Experimental): Designed to train participants in a number of experiential exercises evoking qualities of mindfulness: mental focus, sustained attention and personal and situational awareness. These exercises include versions of the body scan (body awareness exercise), sitting meditation, mindful movement, walking meditation, eating meditation, mindful martial arts exercises and other elements of mindfulness.
  Interventions: Behavioral: Mindfulness-Based Resilience Training

INTERVENTIONS:
Behavioral: Mindfulness-Based Resilience Training — 2.5-day intensive MBRT training sessions.

SUMMARY:
First responders (law enforcement, firefighters, and emergency medical system personnel) are subjected to daily pressures from their duties with resultant compassion fatigue, burnout, anger, poor mental and physical health, maladaptive behavior, and sleep disturbance. The unprecedented heroin and opioid epidemic in West Virginia has accelerated the stresses as these first responders witness overdoses and overdose death on a frequent basis. The plight and suffering of children of the overdose victims is an additional overlooked element in the stress on the first responder community. The proposed project will deliver mindfulness-based resilience training to improve the mental and physical wellbeing, prevent compassion fatigue, burnout, and attrition of first responders and performance improvement by reducing predictable cognitive errors in the Charleston and Huntington areas and measure the effects of this training on this population using validated questionnaires and salivary cortisol before and after the training.

DETAILED DESCRIPTION:
West Virginia (WV) is in the midst of an unprecedented opioid and heroin epidemic with profound social, health, and economic consequences. This stress, especially among law enforcement officials (LEOs), is often experienced within a context of excessive anger, which decreases wellbeing and has the potential to negatively impact public wellbeing as well. These public safety personnel are often left to manage stress and anger in a cultural context that does not support help-seeking behavior and that encourages maladaptive coping mechanisms. Mindfulness-Based Resilience Training (MBRT) has demonstrated significant improvement in self-reported mindfulness, resilience, perceived operational and administrative stress, burnout, emotional intelligence, emotion regulation, mental and physical health, anger, fatigue, and sleep disturbance Introducing effective evidence-based training to first responders has the potential to improve well-being and decrease burnout and improve the performance of the people who protect the community. Should this hypotheses be confirmed, first responders in West Virginia will have an effective intervention to improve resilience, address perceived stress and burnout, and lead to greater mental and physical wellbeing in the face of unprecedented stresses associated with the opioid and heroin epidemic. This would enable this intervention to be scaled across the state among other populations of first responders in this unprecedented public health crisis.

First responders will be recruited from volunteers targeting leadership and thought leaders at the frontline from the three-county area, but primarily from the cities of Charleston and Huntington, to participate in one of two 2.5-day intensive MBRT training sessions. Each 2.5-day session will be coordinated with each agency to ensure maximum participation without disrupting work schedules. Up to 35 participants will participate in each cohort. This study aims to recruit 2 cohorts from the pool of first responders in the Cabell, Kanawha, and Putnam Counties area for a minimum of 50 participants and maximum of 70 participants. Self report measures will be conducted at time 0 (before the intervention), time 1 (after the 2.5-day intensive training), time 2 (4 weeks after the 2.5-day intensive training and after the week 4 remote/virtual booster training) and at time 3 (90 days after the initial intensive training).

ELIGIBILITY:
Inclusion Criteria:

* Current employment as a first responder
* West Virginia residency
* Availability/willingness to engage in a 2.5-day retreat style intervention on identified dates.

Exclusion Criteria:

* Not an actively employed first responder
* Does not currently reside in WV
* Not willing or able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Zullig, PhD, Principal Investigator — West Virginia University
Locations (4):
- United States (4):
  - Kanawha-Charleston Health Department, Charleston, West Virginia
  - Saint John XXIII Pastoral Center, Charleston, West Virginia
  - Marshall University, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No subjects were excluded before assignment. Subjects lost 2 follow up were lost at varying times throughout the 2.5 day period. Mostly due to not showing up for the 2nd and 3rd dates.
Period: Overall Study
Arm/Group | Mindfulness-Based Resilience Training
Started | 30
Completed | 18
Not Completed | 12
Not completed — Withdrawal by Subject | 12

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: The Five Factor Mindfulness Questionnaire (FFMQ). It examines 5 key domains of mindfulness: observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience. Scores range from 39 to 195, with higher scores indicating greater tendency to be mindful.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 111.6 (13.2)

2. Primary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: as for outcome 1
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 115.5 (12.8)

3. Primary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: as for outcome 1
Time Frame: 30 days post intervention
Population: 10 subjects lost to follow up from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 115.3 (10.1)

4. Primary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: as for outcome 1
Time Frame: 90 days post intervention
Population: 12 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 115.6 (12.5)

5. Primary Outcome: Mindfulness Process Questionnaire (MPQ)
Description: The Mindfulness Process Questionnaire (MPQ) is an 8-item self-report measure that assesses the degree to which mindfulness is intentionally practiced or attempted and the ability to bring compassionate awareness to the present moment after observing the attention has drifted off or become judgmental. Items are scored on a Likert type scale ranging from "not at all characteristic of me" to "entirely characteristic of me," and total scores range from 8 to 40, with higher scores indicating greater engagement in mindfulness practices and skills.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 23.4 (4.9)

6. Primary Outcome: Mindfulness Process Questionnaire (MPQ)
Description: as for outcome 5
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 24.8 (14.1)

7. Primary Outcome: Mindfulness Process Questionnaire (MPQ)
Description: as for outcome 5
Time Frame: 30 days post intervention
Population: 10 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 25.5 (3.6)

8. Primary Outcome: Mindfulness Process Questionnaire (MPQ)
Description: as for outcome 5
Time Frame: 90 days post intervention
Population: 12 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 25.7 (4.1)

9. Primary Outcome: Organizational Police Stress Questionnaire
Description: The Police Stress Questionnaire (PSQ) (organizational [OPSQ]) is a 40-item questionnaire consisting of 2 subscales measuring operational stressors (20 job content items) and organizational stressors (20 job context items) on a Likert-type scale, ranging from 1 (no stress at all) to 7 (a lot of stress) and resulting in a maximum score of 140; higher scores indicate greater stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 66.9 (24.8)

10. Primary Outcome: Organizational Police Stress Questionnaire
Description: as for outcome 9
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 64.1 (25.0)

11. Primary Outcome: Organizational Police Stress Questionnaire
Description: as for outcome 9
Time Frame: 30 days post intervention
Population: 10 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 53.4 (22.7)

12. Primary Outcome: Organizational Police Stress Questionnaire
Description: as for outcome 9
Time Frame: 90 days post intervention
Population: 12 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 57.6 (27.6)

13. Primary Outcome: Operational Police Stress Questionnaire
Description: The Police Stress Questionnaire (PSQ) (Operational) is a 40-item questionnaire consisting of 2 subscales measuring operational stressors (20 job content items) and organizational stressors (20 job context items) on a Likert-type scale, ranging from 1 (no stress at all) to 7 (a lot of stress) and resulting in a maximum score of 140; higher scores indicate greater stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 65.3 (27.0)

14. Primary Outcome: Operational Police Stress Questionnaire
Description: as for outcome 13
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 60.5 (19.6)

15. Primary Outcome: Operational Police Stress Questionnaire
Description: as for outcome 13
Time Frame: 30 days post intervention
Population: 10 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 50.6 (18.3)

16. Primary Outcome: Operational Police Stress Questionnaire
Description: as for outcome 13
Time Frame: 90 days post intervention
Population: 12 subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 52.3 (24.9)

17. Primary Outcome: Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale-4 (PSS) is a 4-item scale used to assess perceived stress in life situations. Responses are on a Likert-type scale ranging from "never" to "very often;" higher scores indicate greater perceived stress, with a minimum score of 0 and maximum score of 16.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 8.5 (1.5)

18. Primary Outcome: Perceived Stress Scale (PSS)
Description: as for outcome 17
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 9.2 (1.1)

19. Primary Outcome: Perceived Stress Scale (PSS)
Description: as for outcome 17
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 9.5 (1.5)

20. Primary Outcome: Perceived Stress Scale (PSS)
Description: as for outcome 17
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 8.8 (1.5)

21. Primary Outcome: Emotional Regulation
Description: The Difficulties in Emotional Regulation Scale (DERS) is a 36-item measure that assesses clinically relevant difficulties in emotion regulation. Items range from 1 ("almost never") to 5 ("almost always), and the total score ranges from 36 to 180. Higher scores indicate greater difficulties with emotion regulation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 84.4 (14.4)

22. Primary Outcome: Emotional Regulation
Description: as for outcome 21
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 87.0 (16.9)

23. Primary Outcome: Emotional Regulation
Description: as for outcome 21
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 83.5 (11.0)

24. Primary Outcome: Emotional Regulation
Description: as for outcome 21
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 77.8 (8.5)

25. Primary Outcome: Emotional Intelligence Scale
Description: The Emotional Intelligence Scale (EIS) is a 33-item scale of emotional intelligence. Items are rated on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), and 3 items are reverse scored, producing a score range from 33 to 165. All items are summed to create a total score, and higher scores indicate greater emotional intelligence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 115.5 (11.8)

26. Primary Outcome: Emotional Intelligence Scale
Description: as for outcome 25
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 116.0 (9.9)

27. Primary Outcome: Emotional Intelligence Scale
Description: as for outcome 25
Time Frame: 30 day post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 119.8 (9.9)

28. Primary Outcome: Emotional Intelligence Scale
Description: as for outcome 25
Time Frame: 90 days
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 120.6 (11.5)

29. Primary Outcome: Brief Resilience Scale
Description: The Brief Resilience Scale (BRS) is a 6-item scale designed to assess the ability to recover from stress using a Likert scale, ranging from 1 ("strongly disagree") to 5 (strongly agree). Scores are summed, then divided by the total number of items, to produce a total score ranging from 1 to 5. Higher scores indicate greater resilience.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 2.9 (0.3)

30. Primary Outcome: Brief Resilience Scale
Description: as for outcome 29
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 2.9 (0.3)

31. Primary Outcome: Brief Resilience Scale
Description: as for outcome 29
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 3.0 (0.3)

32. Primary Outcome: Brief Resilience Scale
Description: as for outcome 29
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 3.0 (.2)

33. Primary Outcome: General Family Functioning
Description: The General Family Functioning Subscale (GFF) consists of 12 items. Respondents complete 12 items with a four-point response scale (1 = strongly agree, 4 = strongly disagree). A mean score is computed. Higher scores on the GFF indicate more problematic family functioning. The minimum score on the GFF is 12, and the maximum score is 48.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 34.6 (5.5)

34. Primary Outcome: General Family Functioning
Description: as for outcome 33
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 33.5 (5.6)

35. Primary Outcome: General Family Functioning
Description: as for outcome 33
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 35.8 (1.9)

36. Primary Outcome: General Family Functioning
Description: as for outcome 33
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 35.8 (1.9)

37. Primary Outcome: PROMIS Sleep
Description: Patient Reported Outcomes Measurement Information System (PROMIS®) is comprised of Sleep. Item is rated on a Likert type scale (Score range of 4-19) with higher scores indicating greater symptom severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 11.0 (2.0)

38. Primary Outcome: PROMIS Sleep
Description: as for outcome 37
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 11.1 (1.7)

39. Primary Outcome: PROMIS Sleep
Description: as for outcome 37
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 11.0 (1.3)

40. Primary Outcome: PROMIS Sleep
Description: as for outcome 37
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 10.9 (.9)

41. Primary Outcome: PROMIS Health
Description: Patient Reported Outcomes Measurement Information System (PROMIS®) is comprised of Health. Item is rated on a Likert type scale (Score Range 0-40) with higher scores indicating greater symptom severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 32.5 (4.1)

42. Primary Outcome: PROMIS Health
Description: as for outcome 41
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 32.5 (3.7)

43. Primary Outcome: PROMIS Health
Description: as for outcome 41
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 33.1 (3.8)

44. Primary Outcome: PROMIS Health
Description: as for outcome 41
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 33.3 (4.1)

45. Primary Outcome: PROMIS Fatigue
Description: Patient Reported Outcomes Measurement Information System (PROMIS®) is comprised of Fatigue. Item is rated on a Likert type scale (score range 4-20) with higher scores indicating greater symptom severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 10.9 (2.5)

46. Primary Outcome: PROMIS Fatigue
Description: as for outcome 45
Time Frame: Immediately following intervention
Population: 7 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 11.0 (3.2)

47. Primary Outcome: PROMIS Fatigue
Description: as for outcome 45
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 9.8 (2.6)

48. Primary Outcome: PROMIS Fatigue
Description: as for outcome 45
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 8.9 (2.3)

49. Primary Outcome: PROMIS Anger
Description: Patient Reported Outcomes Measurement Information System (PROMIS®) is comprised of Anger. Item is rated on a Likert type scale (score range 5-25) with higher scores indicating greater symptom severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 30
score on a scale | 13.3 (4.5)

50. Primary Outcome: PROMIS Anger
Description: as for outcome 49
Time Frame: Immediately following intervention
Population: 7 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 23
score on a scale | 12.1 (4.3)

51. Primary Outcome: PROMIS Anger
Description: as for outcome 49
Time Frame: 30 days post intervention
Population: 10 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 20
score on a scale | 11.3 (2.5)

52. Primary Outcome: PROMIS Anger
Description: as for outcome 49
Time Frame: 90 days post intervention
Population: 12 Subjects lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training
Number analyzed (Participants) | 18
score on a scale | 11.3 (2.8)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Mindfulness-Based Resilience Training
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT04929613/Prot_SAP_000.pdf